CLINICAL TRIAL: NCT05463367
Title: Project 1 Aim 2, Adaptations of the Brain in Chronic Pain With Opioid Exposure
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00209670
Record Dates: First submitted 2020-02-27; First posted 2022-07-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use; Opioid Dependence; Opioid-use Disorder; Narcotic Use; Back Pain; Back Injuries; Chronic Pain; Chronic Low-back Pain; Pain, Chronic; Pain;Back Low;Chronic; Pain, Back
Keywords: norco; opioid; pain medication; tramadol; oxycodone; pain; chronic pain; chronic back pain; back pain; narcotics
MeSH Terms: conditions — Opioid-Related Disorders; Back Pain; Back Injuries; Chronic Pain; Pain | interventions — carbidopa, levodopa drug combination; Naproxen; Analgesics, Opioid; oxycodone-acetaminophen; Oxycodone; Oxymorphone; Morphine; Codeine; Tramadol

STUDY DESIGN:
Intervention Model Description: There will be 2 arms of participants, those who have back pain with opioid exposure, and those who have back pain with opioid exposure and opioid misuse disorder. Each participant, regardless of the arm that they are in, will receive each of the possible study interventions. The only difference will be the order of which they receive each interventions.
  Recruitment is completed. Of the collected subjects with opioid exposure none exhibited opioid misuse.
Who Masked: Participant, Investigator
Masking Description: All data analysis personnel are masked regarding groupings
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chronic Back Pain with Opioid Use (Experimental): Subjects of this arms will be on a previously prescribed, short term acting opioid. Previous to each of the three imaging visits, subjects will be instructed to withhold from taking their regular morning opioid dose. Subjects will be randomized into a group that determines the sequence of which they will receive the study drugs. The three sequences are as follows:
  1. treatment dose #1: 25mg carbidopa/ 100mg levodopa + 500mg naproxen, treatment dose #2: subjects prescribed, short acting opioid;
  2. treatment dose #1: placebo, treatment dose #2: subjects prescribed, short acting opioid; or
  3. treatment #1: subjects prescribed, short acting opioid, treatment dose #2: placebo.
  Interventions: Drug: Carbidopa-Levodopa 25 Mg-100 Mg Oral Tablet; Drug: Naproxen 500 Mg; Drug: Opioids
- Chronic Back Pain with Opioid Misuse Disorder (Experimental): Subjects of this arms will be on a previously prescribed, short term acting opioid. Previous to each of the three imaging visits, subjects will be instructed to withhold from taking their regular morning opioid dose. Subjects will be randomized into a group that determines the sequence of which they will receive the study drugs. The three sequences are as follows:
  1. treatment dose #1: 25mg carbidopa/ 100mg levodopa + 500mg naproxen, treatment dose #2: subjects prescribed, short acting opioid;
  2. treatment dose #1: placebo, treatment dose #2: subjects prescribed, short acting opioid; or
  3. treatment #1: subjects prescribed, short acting opioid, treatment dose #2: placebo.
  Interventions: Drug: Carbidopa-Levodopa 25 Mg-100 Mg Oral Tablet; Drug: Naproxen 500 Mg; Drug: Opioids

INTERVENTIONS:
Drug: Carbidopa-Levodopa 25 Mg-100 Mg Oral Tablet — Subjects will receive a single dose of carbidopa/levodopa, when applicable.This will be double-blinded, as neither participants nor study staff will know what medication the participant is receiving.
  Other Names: Sinemet
Drug: Naproxen 500 Mg — Subjects will receive a single dose of naproxen 500mg alongside carbidopa/levodopa, when applicable.This will be double-blinded, as neither participants nor study staff will know what medication the participant is receiving.
  Other Names: Aleve; Anaprox; Antalgin; Midol Extended Relief; Naprosyn; Soproxen; Synflex; Xenobid
Drug: Opioids — Subjects will be pre-screened in regards to their opioid medication. They will receive a single dose of their opioid dose, when appropriate. This will be double-blinded, as neither participants nor study staff will know what medication the participant is receiving.
  Other Names: hydrocodone/acetaminophen; oxycodone/acetaminophen; oxycodone; oxymorphone; morphine; codeine; tramadol

SUMMARY:
This study is designed to track brain functional changes in individuals with i) chronic back pain + opioid use (CBP+O) and individuals with ii) chronic back pain + opioid misuse disorder (CBP+mOUD) following a brief drug delay and re-exposure manipulation. Re-exposure could be placebo, the participant's own opioid dose, or a dopaminergic treatment (DA+NSAID). The participants will be also evaluated for changes in cognition, emotion, and motor abilities with opioid delay and re-exposure to placebo, opioid, or DA+NSAID.

DETAILED DESCRIPTION:
Screening Visit (2-3 hours) (if applicable):

Participants that have participated in Project 1 Aim 1 within three months of consenting to Project 1 Aim 2 will not require a screening visit and can continue on to Visit 1, 2 and 3 of Aim 2.

A screening visit will be applicable for those participants that did not participate in Project 1 Aim 1, and for those that had participated but did so more than three months prior to consenting to Project 1 Aim 2.

Participants will be evaluated with inclusion/exclusion criteria and complete the informed consent. A medical/pain history will be taken and a physical exam will be completed by a physician. Participants will complete a number of questionnaires assessing health and medical history, past and current pain levels, and personality. Participants will have their blood drawn to confirm appropriate kidney and liver function (investigators will take ~40mL of blood). Participants will also be asked to provide a urine sample to confirm if any illicit drugs are in their system.

Participants will also be instructed to report their pain and craving ratings via an application that will be downloaded on their device. They will need to complete two ratings per day that they are involved in the study.

Visit 1, 2, and 3 (6-8 hours):

Participants will be instructed to not take their morning opioid medication. Upon arrival, participants will be asked to report their pain and craving using the Pain and Craving Index (PCI), which will be used as a baseline rating. They will complete the PCI once every hour throughout their visit. Once their PCI has increased by at least two-points from their baseline rating, the patient will undergo their first brain MRI scan (anatomical and functional scans).

Between arrival and the first MRI, participants will complete several questionnaires regarding pain, mood, thoughts, and feelings. Directly after the MRI, participants will have their blood drawn. This blood draw will be used to quantitatively analyze the participants' opioid levels. Participants will then complete the NIH Toolbox. The NIH Toolbox is a compilation of activities that evaluate different cognitive, motor and emotional functions.

Participants will then be randomized and receive "Treatment Dose #1." Treatment dose #1 will be one of the following: a single dose of the participant's opioid prescription (provided by Northwestern Memorial Hospital's investigational pharmacy), carbidopa/levodopa (c-dopa/l-dopa), or placebo (lactose). Participants will then complete the same questionnaires as they previously had, undergo a second brain MRI scan, have their blood drawn, and complete a second NIH Toolbox.

Participants will then receive "Treatment Dose #2." For those participants that received their opioid medication for treatment dose #1, they will receive placebo for their treatment dose #2. For those participants that received carbidopa/levodopa or placebo for treatment dose #1, they will receive their opioid prescription for their treatment dose #2.

After receiving treatment dose #2, participants will be done with their imaging visit.

Each participant will have three total imaging visits. The activities within each imaging visit will be identical, the only variable will be the study intervention (opioid, c-dopa/l-dopa, or placebo) that they receive. All participants will receive each of the possible study interventions; however, the sequence of when they will receive each drug will be different from participant to participant. Neither participants nor the clinical coordinator/assistant will know which intervention the participant is receiving.

ELIGIBILITY:
Inclusion Criteria:

* History of low back pain for a minimum of 6 months daily (prior to screening), meeting the Quebec Task Force Classification System symptom categories I-III;
* Male or female, age equal or greater than 18 years, with no racial/ethnic restrictions;
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires;
* Must be in generally stable health;
* Must sign an informed consent document after a complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits and potential risks, and are willing to participate;
* Must have, on average ≥ 4/10 units of pain intensity over the course of a 1-4 week period prior to the brain scanning visit;
* Must be willing to complete daily smartphone/computer eDiary ratings;
* Must be on regular opioid therapy or for at least 3 months prior to randomization which will be up to the clinical investigator's decision
* Must be on a short acting opioid therapy (anticipated duration of action < 6 hours)

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills;
* Other comorbid chronic pain or neurological conditions;
* Use of therapeutic doses of antidepressant medications at unstable doses (i.e., tricyclic depressants, SSRIs, SNRIs; low doses used for sleep may be allowed);
* Significant other unstable medical disease such as diabetes, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy;
* Uncontrolled hypertension;
* Renal insufficiency;(correlated creatinine clearance < 40mL/min or serum creatinine ≥2)
* Daily use of high doses of opioids,, as defined as > 50mg morphine equivalent/day;
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Evidence of poor treatment compliance, in the judgment of the investigator;
* Intra-axial implants (e.g. spinal cord stimulators or pumps);
* All exclusion criteria for MR safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia;
* Pregnancy, or inability to use an effective form of contraception in women of child-bearing age;
* An established diagnosis of diabetes (type 1 or type 2)
* Lactose intolerance
* History of an allergic reaction to naproxen or any NSAID;
* History of any untoward reaction to carbidopa/levodopa
* Use of a patch or long acting opioid therapy (e.g. anticipated duration of action > 6 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences across drugs in Withdrawal relief assessed by Pain and Craving Index (PCI). | 3 weeks
  Pain and Drug craving Index (PCI) will be used to evaluate self-reported medication cravings. Participants will complete the scale, before and after receiving the visit drug treatment. Changes in PCI scores (after minus before) will be compared between drugs (opioids vs. placebo vs. Carbidopa/Levodopa +naproxen).
Differences across drugs in pain changes as assessed by Numeric Rating Scale (0-10). | 3 weeks
  NRS scale will be used to evaluate self-reported pain. Participants will rate their pain before and after receiving the visit drug treatment. Changes in pain scores (after minus before) will be compared between drugs (opioids vs. placebo vs. Carbidopa/Levodopa +naproxen).

SECONDARY OUTCOMES:
Differences in pain changes (NRS) across High and Low Misuse groups measured by the Current Opioid Misuse Measure (COMM). | 3 weeks
  Current Opioid Misuse Measure (COMM) is a 17-item self-report measure of risk for aberrant medication-related behavior among persons with chronic pain who are prescribed opioids for pain. Participants will be divided into two groups: high COMM and low COMM. Changes in pain scores (after minus before) will be compared between COMM groups (high vs. low)
Differences in withdrawal changes (PCI) across High and Low Misuse groups measured by the Current Opioid Misuse Measure (COMM). | 3 weeks
  Current Opioid Misuse Measure (COMM) is a 17-item self-report measure of risk for aberrant medication-related behavior among persons with chronic pain who are prescribed opioids for pain. Participants will be divided into two groups: high COMM and low COMM. Changes in Withdrawal relief - PCI score (after minus before) will be compared between COMM groups (high vs. low).
Whole-cortex multi-receptor related activity | 3 weeks
  We used the resting-state fMRI to generate whole-brain voxel-wise amplitude of low-frequency fluctuations (ALFF) maps that reflect the low-frequency energy of spontaneous BOLD activity. Cortex-wide receptor-related activity for each subject will be computed as the normalized dot product between ALFF maps and the standardized receptor density distribution maps obtained from Hensen et al 2022. This will result in one value per subject representing cortical receptor-related activity for any given receptor type. For this analysis we will focus on 3 receptors that we have shown to be modulated in long-term opioid use including the serotonin (5-HT1A and 5-HT1B) receptors and the µ-opioid (MOR) receptor. We will also investigate both dopamine (D1 and D2) receptors to test their modulation with administering dopamine+NSAID.

CONTACTS AND LOCATIONS:
Overall Officials: Apkar V Apkarian, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

DOCUMENTS (2):
  • Study Protocol (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05463367/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT05463367/SAP_001.pdf